CLINICAL TRIAL: NCT04257643
Title: Efficacy of Aquatic Based Versus Land-based Exercise in Lymph Edema Post-mastectomy: a Prospective Randomized Controlled Trial.
Brief Title: Aquatic Versus Land Based Exercise on Lymphedema Post Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadaya Mosaad, Principal investigator., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/002615
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: Aquatic exercise-; Land based exercise; lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): water-based exercise was conducted at a hydrotherapy pool for the Eden Heelth Care,Cairo The pool measures 8 × 15 m and ranges from 1 to 1.8 m in depth with access via steps. Interventions were conducted predominately in the deeper section of the pool so participants immerse their neck in water. Thermo neutral water temperature, 30-32 °C at room temperature. Females were instructed to adjust water depth completely covering clavicles from standing position. Diaphragmatic breathing during exercise routine to assist with lymph fluid clearance. Exercise continuously for 40 to 45 min Full-body warm-up exercise for 10 min and cooling down for 10 minutes. Plus land-based exercise session for 60 minutes for 8 weeks in the form of warm-up, strengthening, and cooling down exercise.
  Interventions: Other: aquatic based exercise.; Other: land-based exercise.
- Control group (Active Comparator): Land-based exercise program: Supervised program consisted of 60-min sessions, three times a week, over 8 weeks. The exercise program consisted of the first 10 minutes for warm-up exercise with a small softball, fit -ball, mobility and stretching exercise. Then 30-40 minutes for strength development with different materials and positions, that require more body control and increase joint motion. Then the last 10 minutes for cooling down for stretching exercise for the arm muscles
  Interventions: Other: land-based exercise.

INTERVENTIONS:
Other: aquatic based exercise. — exercise under water with the patient standing in a swimming pool, for 60 minswith water to the neck and then practice the arm exercise plus the diaphragmatic breathing exercise. The duration of the exercise programs was selected to be 60 minutes, 3 days per week for 8-week intervention
  Arms: Experimental group
Other: land-based exercise. — land-based exercise session for 60 minutes for 8 weeks in the form of warm-up, strengthening, and cooling down exercise.Land-based exercise program: Supervised program consisted of 60-min sessions, three times a week, over 8 weeks. The exercise program consisted of the first 10 minutes for warm-up exercise with a small softball, fit -ball, mobility and stretching exercise. Then 30-40 minutes for strength development with different materials and positions, that require more body control and increase joint motion. Then the last 10 minutes for cooling down for stretching exercise for the arm muscles [14]. Women were asked to exercise continuously for 60 mins, by performing the arm exercises by repeating the session, and were instructed to exercise at moderate intensity .

SUMMARY:
Fifty eligible breast cancer survivors (median, 10 yrs after surgery) with arm lymph-edema (median, 21% inter limb difference) were included and randomized into the intervention(group A, n = 25) or control ( Group B, n = 25). Intervention group received 60 minutes aquatic-based exercise in the form of warm-up for 10 mins, then strengthening exercise for 40 minutes, followed by 10 min cooling down in the form of stretching and mobility exercise, three times a week for 8 weeks, plus land-based exercise session for 60 minutes for 8 weeks in the form of warm-up, strengthening, and cooling down exercise. The control group received 60 minutes of land base exercise, three times a week, for 8 weeks. Arm volume, shoulder flexion, abduction range of motion and pain using a visual analogue scale were assessed at baseline and after 8 weeks of treatment.

DETAILED DESCRIPTION:
Group A: 25 female Patients there aged ranged from 37 to 67 years old with BCRL, in Group-A had been dealt with water-based exercise was conducted at a hydrotherapy pool for the Eden Health care, cairo, The pool measures 8 × 15 m and ranges from 1 to 1.8 m in depth with access via steps. Interventions were conducted predominately in the deeper section of the pool so participants immerse their neck in water.

Control group, Group B: 25 female Patients there aged ranged from 37 to 67 years old with BCRL, in control group had been dealt Land-based exercise program: Supervised program consisted of 60-min sessions, three times a week, over 8 weeks. The exercise program consisted of the first 10 minutes for warm-up exercise with a small softball, fit -ball, mobility and stretching exercise. Then 30-40 minutes for strength development with different materials and positions, that require more body control and increase joint motion. Then the last 10 minutes for cooling down for stretching exercise for the arm muscles .

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer with unilateral axillary lymph node excision.
* Mild-moderate degreed lymphedema (stage I and II) .
* Lymphedema with a duration of at least 1 year .

Exclusion Criteria:

* Recurrence of cancer.
* Ongoing active oncological treatment.
* Functional disorders hindering participation in exercise programs.
* Open wound at any area of the body.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Limb volume measurement: | 8 weeks.
  the patient in a comfortable sitting position, a standard one cm, retractable, the fibreglass tape measure was used to perform circumference measurement. The measurement was made at, 10, 20, 30, and 40 cm above the ulnar styloid process,

SECONDARY OUTCOMES:
Range of Motion | 8 weeks.
  Upper extremity active ROM for shoulder flexion and abduction were assessed in the standing position using a standard goniometric method

OTHER OUTCOMES:
Visual analogue scale for pain assessment | 8 weeks.
  horizontal (HVAS) or vertical (VVAS) line, usually 10 centimetres (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. Instructions, the time period for reporting, and verbal descriptor anchors have varied widely in the literature depending on the intended use of the scale

CONTACTS AND LOCATIONS:
Overall Officials: Khadra M Ali, Phd, Principal Investigator — Cairo University, Faculty of physical Therapy.
Locations (1):
- Cairo university., Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP
Time Frame: We will share results after 6 months from publication.